CLINICAL TRIAL: NCT01236014
Title: Indirect Comparison of Efficacy of Treatments for Idiopathic Immune Thrombocytopenic Purpura - Review of Platelet Responses and Bleeding Events
Brief Title: Indirect Comparison Between Eltrombopag & Romiplostim
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 114014
Record Dates: First submitted 2010-11-04; First posted 2010-11-08 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Thrombocytopaenia
MeSH Terms: conditions — Thrombocytopenia | interventions — eltrombopag; romiplostim

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Eltrombopag & standard of care
  Interventions: Drug: Eltrombopag
- Romiplostim & standard of care
  Interventions: Drug: Romiplostim
- Standard of care
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eltrombopag — Eltrombopag & standard of care
  Groups: Eltrombopag & standard of care
Drug: Romiplostim — Romiplostim & standard of care
  Groups: Romiplostim & standard of care
Drug: Placebo — Placebo & standard of care
  Groups: Standard of care

SUMMARY:
An indirect comparison to compare the efficacy of eltrombopag versus romiplostim

DETAILED DESCRIPTION:
An indirect analysis was conducted to evaluate the relative efficacy of eltrombopag and romiplostim using placebo as a common comparator

ELIGIBILITY:
Inclusion Criteria:

* Adults with ITP
* Pre-specified treatment
* Prospective clinical studies with at least 10 patients

Exclusion Criteria:

* Adults with ITP for other reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Identified through a systematic review: TRA102537, Kuter 2008
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2009-08; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Durable response: platelet count of >=50 and <400 Gi/L | 6 months
Overall response: either a durable response or a transient platelet response | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline